CLINICAL TRIAL: NCT05357742
Title: Basic Needs Navigation Intervention to Address Multidimensional Adversity in African Americans With Diabetic Kidney Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Mukoso N. Ozieh, Assistant Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: PRO00041675; R21DK131356 (NIH)
Record Dates: First submitted 2022-04-27; First posted 2022-05-03 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Diabetic Nephropathies; Diabetes Mellitus, Type 2; Chronic Kidney Diseases; Healthy Lifestyle
Keywords: Social risk factors; Social determinants of health
MeSH Terms: conditions — Diabetic Nephropathies; Diabetes Mellitus, Type 2; Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants randomized to the intervention group will receive the manualized study intervention delivered by a health educator via telephone weekly for 12-weeks, followed by three monthly booster sessions resulting in a total of 6 months intervention.
  Interventions: Behavioral: Individualized basic need navigation and lifestyle coaching and skills training
- Control group (Active Comparator): Participants randomized to the control group will receive the manualized study intervention delivered by a health educator via telephone weekly for 12-weeks, followed by three monthly booster sessions resulting in a total of 6 months intervention.
  Interventions: Behavioral: Enhanced usual care

INTERVENTIONS:
Behavioral: Individualized basic need navigation and lifestyle coaching and skills training — During each session participants will receive the manualized study intervention which includes 1) DKD education, 2) Individualized basic needs navigation, and 3) Lifestyle coaching and skills training. Participants will be provided a FORA 2-in-1 device with glucose test strips to allow testing at least once a day. The device automatically uploads blood pressure and glucose readings to a secure server in real time and the health educator will have access to this secure server. Readings will be used to guide lifestyle coaching and skills training.
  Arms: Intervention Group
Behavioral: Enhanced usual care — During each session participants will receive DKD education only.
  Arms: Control group

SUMMARY:
The overarching goal of this proposal is to test the feasibility of a basic needs navigation intervention on improving clinical outcomes, self-care behaviors and quality of life in low-income African Americans with diabetic kidney disease (DKD) experiencing multidimensional adversity.

The study objective will be achieved with the following aims:

Aim 1: To determine the feasibility of a basic needs navigation intervention as measured by recruitment, session attendance and retention in low-income Africans Americans with DKD experiencing multidimensional adversity.

Aim 2: To determine the frequency and compounding nature of different basic needs in Africans Americans with DKD experiencing multidimensional adversity to help refine the basic needs navigation intervention.

Aim 3: To evaluate the change and variability in the clinical outcomes (hemoglobin A1c, blood pressure, lipids) at 6 months of follow-up to plan for larger trial.

DETAILED DESCRIPTION:
Multidimensional adversity, defined as having three or more social adversities such as housing instability, food insecurity, transportation needs, utility needs, interpersonal safety, and financial strain impacts the complex self-management of DKD and negatively impacts health outcomes. Evidence suggests patient navigation programs may be a promising strategy to improve health outcomes in low-income individuals with chronic disease. However, there is limited evidence on the use of patient navigator programs to address multidimensional adversity in individuals with chronic disease. Therefore, the primary objective of this study is to address this gap in knowledge.

Study overview: This will be accomplished using a two-arm pilot randomized control trial. Fifty (50) African American adults with DKD experiencing multidimensional adversity will be randomized into one of two arms: 1) Intervention arm and 2) Enhanced usual care arm.

Description of intervention: Participants randomized to the intervention arm will receive the manualized study intervention which includes three components 1) DKD education, 2) Individualized basic needs navigation, and 3) Lifestyle coaching and skills training. Participants will be provided a FORA 2-in-1 device with glucose test strips to allow testing at least once a day. The device automatically uploads blood pressure and glucose readings to a secure server in real time and the health educator will have access to this secure server. Readings will be used to guide lifestyle coaching and skills training. All participants will be assessed at baseline, 3- and 6-months for clinical outcomes (hemoglobin A1c, blood pressure, lipids), self-care behaviors (diet, exercise, and medication adherence), and quality of life (SF-12).

Control arm (Enhanced usual care arm): Participants randomized to the control arm will receive the manualized study intervention which incudes only DKD education.

All participants will be assessed at baseline, 3- and 6-months for clinical outcomes (hemoglobin A1c, blood pressure, lipids), self-care behaviors (diet, exercise, and medication adherence), and quality of life (SF-12).

ELIGIBILITY:
Inclusion Criteria:

1. self- report as Black/African American
2. age ≥18
3. screen positive for 1 or more adversities using the Centers for Medicare and Medicaid Services Accountable Health Communities Health-Related Social Needs Screening tool
4. diagnosed type 2 diabetes (T2DM) with HbA1c≥8
5. chronic kidney disease (CKD)
6. able to communicate in English.

Exclusion Criteria:

1. does not identify as Black/African American
2. age <18
3. no diagnosis of T2DM and CKD
4. cognitive impairment at screening visit
5. active psychosis
6. active alcohol or drug abuse/dependency
7. life expectancy <12 months
8. participation in other diabetes/CKD trials
9. unable to communicate in English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Feasibility of the basic needs navigation intervention | At 6 months post intervention follow-up
  Feasibility of the basic needs navigation intervention as measured by recruitment, session attendance and retention

SECONDARY OUTCOMES:
Basic Needs | At 6 months post intervention follow-up
  Frequency of basic needs will be assessed using the Centers for Medicare and Medicaid Services Accountable Health Communities Health-Related Social Needs Screening tool
Hemoglobin A1c (Hb A1c) | Change in baseline Hb A1c at 6 months post intervention follow-up
  Blood will be drawn by trained phlebotomist for HbA1c
Systolic blood pressure (SBP) | Change in baseline SBP at 6 months post intervention follow-up
  Blood pressure readings will be obtained using automated BP monitors (OMRON IntelliSenseTM HEM-907XL)
LDL cholesterol | Change in baseline LDL at 6 months post intervention follow-up
  Blood sample will be drawn by a trained phlebotomist and sent to the laboratory for LDL cholesterol.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

REFERENCES:
- [Derived] Ozieh MN, Patterson CG, Williams JS, Walker RJ, Egede LE. Basic needs navigation intervention to address multidimensional adversity in African Americans with diabetic kidney disease: A pilot randomized clinical trial protocol. Contemp Clin Trials. 2025 Dec 17;161:108183. doi: 10.1016/j.cct.2025.108183. Online ahead of print. PMID 41419054